CLINICAL TRIAL: NCT00888550
Title: A Randomized Trial of Post-Operative Outcomes: Splinting Versus Not Splinting of the Distal Lower Extremity After Intramedullary Nailing for Tibial Fractures
Brief Title: Splinting Versus Not Splinting of the Distal Lower Extremity After Intramedullary Nailing for Tibial Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Steven Morgan, MD, Denver Health Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHMC07-0216
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Tibia Fracture
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1. Splinting (Experimental)
  Interventions: Procedure: Post-Op Splinting
- 2. No Splinting (Active Comparator)
  Interventions: Procedure: No Splinting

INTERVENTIONS:
Procedure: Post-Op Splinting — Splint will applied post-operatively and will remain on for two weeks
  Arms: 1. Splinting
Procedure: No Splinting — Patient will be discharged post-operatively without a splint on their lower leg.
  Arms: 2. No Splinting

SUMMARY:
Two standards of care exist with regards to posterior splinting post-operatively. The proponents of splinting feel the additional immobilization decreases the stress on the soft tissue, subsequently preventing or limiting pain while improving early range of motion (ROM). The opposing belief is that the splinting is without therapeutic benefit and that early mobilization is beneficial. With regards to both practices, the surgeon's practice is anecdotally based on past experience.

The purpose of this study is to compare the results obtained with and without posterior splinting after intramedullary (IM) nailing for tibia fractures in order to provide evidence based reasoning to guide future practice.

ELIGIBILITY:
Inclusion Criteria:

* Isolated tibia fracture that is open grade II or less and all closed tibia fractures that are amenable to treatment with an IM nail

Exclusion Criteria:

* Pregnant Women
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Differences across time and between groups for pain and range of motion | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States